CLINICAL TRIAL: NCT04650477
Title: Does Forearm Position Matter in Subpectoral Biceps Tenodesis? A Randomised Controlled Trial
Brief Title: Forearm Position in Subpectoral Biceps Tenodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist,Chief assistant, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Forearm position in tenodesis
Record Dates: First submitted 2020-11-09; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Biceps Tendon Disorder
Keywords: biceps; tenodesis; forearm; shoulder arthroscopy; position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixated in the EP position (Active Comparator): Long head of biceps tenodesis was performed for 25 patients whose joints were fixated while forearm in the extension-pronation (EP) position
  Interventions: Procedure: Fixation while forearm in extension-pronation position
- Fixated in the neutral position (No Intervention): Long head of biceps tenodesis was performed for 25 patients whose joints were fixated while forearm in the neutral position (elbow 90 degrees flexed and hands positioned with the thump pointing up

INTERVENTIONS:
Procedure: Fixation while forearm in extension-pronation position — Fixation was performed after tenodesis in the extension-pronation position, which is the anatomically most suitable position of the biceps tendon.
  Arms: Fixated in the EP position

SUMMARY:
The investigators aimed to compare two different forearm positions, extension-pronation (EP) or neutral, for fixation of the long head of the biceps tendon (LHB) in biceps tenodesis.

DETAILED DESCRIPTION:
Long head of biceps pathologies have been regarded as a source of anterior shoulder pain and disability. Tenodesis is preferable surgical choice for especially young patients to to eliminate anterior shoulder pain. The optimal position of the elbow and forearm during tenodesis is a debated topic. The investigators aimed to evaluate pain and strength loss after biceps tenodesis fixed at extension-pronation (EP) and neutral positions. The investigators aimed to find the most appropriate and anatomical arm position that gives better clinical and functional results.

ELIGIBILITY:
Inclusion Criteria:

-Participants with diagnosis of chronic biceps tendinitis

Exclusion Criteria:

- Participants who had undergone rotator cuff repair surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the two groups in terms of functional score | 6 months
  The investigators evaluated the functional results of the patients with the Ases score. 100 points is the best result in 17 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Karslıoğlu, Study Chair — SBU Prof Cemil Tascioglu City Hospital
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ahrens PM, Boileau P. The long head of biceps and associated tendinopathy. J Bone Joint Surg Br. 2007 Aug;89(8):1001-9. doi: 10.1302/0301-620X.89B8.19278. PMID 17785735
- [Background] Alpantaki K, McLaughlin D, Karagogeos D, Hadjipavlou A, Kontakis G. Sympathetic and sensory neural elements in the tendon of the long head of the biceps. J Bone Joint Surg Am. 2005 Jul;87(7):1580-3. doi: 10.2106/JBJS.D.02840. PMID 15995126
- [Background] Arena C, Dhawan A. Mini-open Subpectoral Biceps Tenodesis Using a Suture Anchor. Arthrosc Tech. 2017 Sep 18;6(5):e1625-e1631. doi: 10.1016/j.eats.2017.06.019. eCollection 2017 Oct. PMID 29399446
- [Background] Baker BE, Bierwagen D. Rupture of the distal tendon of the biceps brachii. Operative versus non-operative treatment. J Bone Joint Surg Am. 1985 Mar;67(3):414-7. PMID 3972865
- [Background] Ball C, Galatz LM, Yamaguchi K. Tenodesis or tenotomy of the biceps tendon: Why and when to do it. Tech Shoulder Elb Surg 2001;2:140-152. doi:10.1097/00132589-200109000-00002
- [Background] Boileau P, Krishnan SG, Coste JS, Walch G. Arthroscopic biceps tenodesis: a new technique using bioabsorbable interference screw fixation. Arthroscopy. 2002 Nov-Dec;18(9):1002-12. doi: 10.1053/jars.2002.36488. PMID 12426544
- [Background] Boileau P, Neyton L. Arthroscopic tenodesis for lesions of the long head of the biceps. Oper Orthop Traumatol. 2005 Dec;17(6):601-23. doi: 10.1007/s00064-005-1154-y. English, German. PMID 16369756
- [Background] Eames MH, Bain GI, Fogg QA, van Riet RP. Distal biceps tendon anatomy: a cadaveric study. J Bone Joint Surg Am. 2007 May;89(5):1044-9. doi: 10.2106/JBJS.D.02992. PMID 17473142
- [Background] Fellows SJ, Rack PM. Changes in the length of the human biceps brachii muscle during elbow movements. J Physiol. 1987 Feb;383:405-12. doi: 10.1113/jphysiol.1987.sp016416. PMID 3656128
- [Background] Fogg QA, Hess BR, Rodgers KG, Ashwood N. Distal biceps brachii tendon anatomy revisited from a surgical perspective. Clin Anat. 2009 Apr;22(3):346-51. doi: 10.1002/ca.20786. PMID 19280656
- [Background] Forman DA, Abdel-Malek D, Bunce CMF, Holmes MWR. Muscle length and joint angle influence spinal but not corticospinal excitability to the biceps brachii across forearm postures. J Neurophysiol. 2019 Jul 1;122(1):413-423. doi: 10.1152/jn.00620.2018. Epub 2019 May 22. PMID 31116661
- [Background] Gill TJ, McIrvin E, Mair SD, Hawkins RJ. Results of biceps tenotomy for treatment of pathology of the long head of the biceps brachii. J Shoulder Elbow Surg. 2001 May-Jun;10(3):247-9. doi: 10.1067/mse.2001.114259. PMID 11408906
- [Background] Itoi E, Kuechle DK, Newman SR, Morrey BF, An KN. Stabilising function of the biceps in stable and unstable shoulders. J Bone Joint Surg Br. 1993 Jul;75(4):546-50. doi: 10.1302/0301-620X.75B4.8331107.
- [Background] Jarrett CD, Weir DM, Stuffmann ES, Jain S, Miller MC, Schmidt CC. Anatomic and biomechanical analysis of the short and long head components of the distal biceps tendon. J Shoulder Elbow Surg. 2012 Jul;21(7):942-8. doi: 10.1016/j.jse.2011.04.030. Epub 2011 Aug 3. PMID 21813298
- [Background] Kilicoglu O, Koyuncu O, Demirhan M, Esenyel CZ, Atalar AC, Ozsoy S, Bozdag E, Sunbuloglu E, Bilgic B. Time-dependent changes in failure loads of 3 biceps tenodesis techniques: in vivo study in a sheep model. Am J Sports Med. 2005 Oct;33(10):1536-44. doi: 10.1177/0363546505274716. Epub 2005 Jul 11. PMID 16009989
- [Background] Kumar VP, Satku K, Balasubramaniam P. The role of the long head of biceps brachii in the stabilization of the head of the humerus. Clin Orthop Relat Res. 1989 Jul;(244):172-5. PMID 2743659
- [Background] Lo IK, Burkhart SS. Arthroscopic biceps tenodesis: Indications and technique. Oper Tech Sports Med 2002;10:105-112. doi:10.1053/otsm.2002.30651
- [Background] Lo IK, Burkhart SS. Arthroscopic biceps tenodesis using a bioabsorbable interference screw. Arthroscopy. 2004 Jan;20(1):85-95. doi: 10.1016/j.arthro.2003.11.017. PMID 14716285
- [Background] Maynou C, Mehdi N, Cassagnaud X, Audebert S, Mestdagh H. [Clinical results of arthroscopic tenotomy of the long head of the biceps brachii in full thickness tears of the rotator cuff without repair: 40 cases]. Rev Chir Orthop Reparatrice Appar Mot. 2005 Jun;91(4):300-6. doi: 10.1016/s0035-1040(05)84327-2. French. PMID 16158544
- [Background] Neviaser AS, Patterson DC, Cagle PJ, Parsons BO, Flatow EL. Anatomic landmarks for arthroscopic suprapectoral biceps tenodesis: a cadaveric study. J Shoulder Elbow Surg. 2018 Jul;27(7):1172-1177. doi: 10.1016/j.jse.2018.01.007. Epub 2018 Feb 27. PMID 29500072
- [Background] Pfahler M, Branner S, Refior HJ. The role of the bicipital groove in tendopathy of the long biceps tendon. J Shoulder Elbow Surg. 1999 Sep-Oct;8(5):419-24. doi: 10.1016/s1058-2746(99)90070-8. PMID 10543593